CLINICAL TRIAL: NCT04043949
Title: The Influences of Dry Eye Disease on Optical Quality
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DEDOQ
Record Dates: First submitted 2018-12-05; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2017-12

CONDITIONS: Dry Eye; Vision; Disturbance, Hysterical
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal: healthy subjects
- Dry eye group: patients with dry eye
- Dry eye after treatment: patients with dry eye after treatment

SUMMARY:
DED could result in visual disturbance and damage optical quality. We aimed to evaluate the influences of dry eye disease (DED) on optical quality and their correlations.

DETAILED DESCRIPTION:
This study is aimed at evaluating changes of optical quality in dry eye patients with superficial punctate keratopathy after being treated by artificial lubricant and anti-inflammatory eye drops.

ELIGIBILITY:
Inclusion Criteria:

1. patients were diagnosed as dry eye according to the criteria provided by the Dry Eye Workshop (DEWS)
2. positive corneal fluorescein staining (CFS)
3. best-corrected distance visual acuity better than 20/20.

Exclusion Criteria:

History of ocular surgeries, contact lens wear, meibomian gland dysfunction, and any type of corneal scarring such as dystrophies or infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged between 18-65 years old.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
The severity of DED influenced the optical quality of dry eye patients | 2017.7-2019.7
  The optical quality of dry eye patients
High order abberations | 2017.7-2019.7
  cornela high order abberations of patients

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, MD,Phd, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided